CLINICAL TRIAL: NCT06802172
Title: Modified Title Project 4: Effect of Meal Timing During Cancer Treatment in Alaska Native Patients: A Randomized Clinical Trial
Brief Title: Modified Title Project 4: Effect of Meal Timing During Cancer Treatment in Alaska Native Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Alaska Native Tribal Health Consortium (Other); Alaska Native Medical Center (Other); Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Timothy Thomas, MD, Director, Research Services, Alaska Native Tribal Health Consortium
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RG1124486; 1P50CA285275-01A1 (NIH); 2111923-7 (Other: Alaska Area Institutional Review Board (AAIRB))
Record Dates: First submitted 2025-01-27; First posted 2025-01-31 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Rectal Cancer Stage II; Rectal Cancer Stage III; Breast Cancer Stage I
Keywords: Time-restricted eating; Time restricted eating; Meal timing
MeSH Terms: conditions — Rectal Neoplasms; Breast Neoplasms; Intermittent Fasting

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Time-restricted eating (TRE) (Experimental): Participants assigned to the TRE group will have an 8-hour daily eating period, starting 1-3 hours after waking up [8 hours eating / 16 hours fasting per day (6+ days a week)].
  Interventions: Behavioral: Time-restricted eating; Other: Questionnaire Administration; Procedure: Biospecimen Collection; Behavioral: Health coaching
- Control group (Active Comparator): Participants assigned to the control group are not time-restricted, and have a 12+ hour window of eating per day.
  Interventions: Other: Questionnaire Administration; Procedure: Biospecimen Collection; Behavioral: Health coaching

INTERVENTIONS:
Behavioral: Time-restricted eating — Participate in time-restricted eating plan
  Arms: Time-restricted eating (TRE)
Other: Questionnaire Administration — Complete questionnaire
Procedure: Biospecimen Collection — Undergo collection of blood and stool
Behavioral: Health coaching — Receive nutrition counseling

SUMMARY:
The goal of this clinical trial is to test meal-timing as a novel and sustainable interventional approach during cancer treatment to improve therapeutic response and metabolic health in an understudied population. This clinical trial will enroll patients with rectal or breast cancer receiving neoadjuvant treatment at the Alaska Native Medical Center (ANMC), which is part of the Alaska Native Tribal Health Consortium (ANTHC).

A promising strategy for improving the efficacy of anticancer treatments and reducing associated toxicities involves combining treatment with fasting regimens. In pre-clinical and clinical studies, various forms of fasting have been shown to induce tumor regression and improve long-term survival. According to the differential stress sensitization theory, fasting is thought to sensitize tumor cells to the cytotoxic effects of chemotherapy and radiation, while protecting healthy cells by increasing stress resistance. While healthy cells slow their growth and become more stress resistant in response to fasting, cancer cells cannot survive in nutrient-deficient environments; although the underlying mechanisms are not fully understood. However, extended water-only fasting can be challenging for patients and poses undue health risks. Intermittent fasting, and specifically time-restricted eating (TRE), may offer a viable alternative. TRE involves eating within a shorter window (e.g., 8 hours) and fasting for the remainder of the day but involves no other dietary restrictions. Because of its simplicity, TRE may be more sustainable than other fasting regimens. TRE also improves several cardio-metabolic endpoints, including insulin sensitivity, which may also be beneficial during anticancer treatments.

DETAILED DESCRIPTION:
Participants will be randomized to one of two groups:

1. Time-restricted eating (TRE) (8-hour daily eating period, starting 1-3 hours after waking up), OR
2. A control group defined as a ≥12-hour daily eating period.

Participants are assigned to either TRE (8-hour daily eating period, starting 1-3 hours after waking up) or a control group defined as a ≥12-hour daily eating period. Their randomized meal assignment arm begins no later than 1-2 week after they begin cancer treatment and ends at end of treatment (resection if indicated). This is a period of approximately 6 months.

During this time, participants will be asked to record the time they started and finished eating every day. Electronic reminders and weekly calls to the participants will be made by study staff who maintain records of patient's meal timing. Researchers will time the TRE schedules relative to sleep time (not time of day), which is a reasonable proxy for circadian time. The control group was designed to mimic typical eating habits in the U.S., as data from NHANES suggest that the median American eats over a 12.5-hour period each day. Aside from these general prescriptions, no set number of snacks, meals, or calories will be prescribed. Instead, researchers will measure how TRE affects self-reported mealtimes, meal frequency, and food intake through a combination of daily adherence surveys, 3-day food records and continuous glucose monitoring (CGM).

Participants will receive weekly one-on-one nutrition counseling during the first month and then monthly counseling sessions thereafter. Participants will complete questionnaires at intake and subsequent follow-up assessments. Blood and stool samples will also be collected from participants throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Self-identify as Alaska Native or American Indian person and eligible for care at the ANMC
* Age≥21 years
* Histologically confirmed rectal cancer stage II,III, or IV (if curative) per AJCC criteria
* Histologically confirmed HER2+ or triple negative breast cancer stage I, II, or III, per AJCC criteria
* BMI≥18.5 kg/m2
* Plan to receive neoadjuvant therapy
* Must have capacity to give informed consent
* Willing and able to adhere to the assessments, visit schedules, prohibitions, and restrictions
* Has completed ≤ 4 weeks of neoadjuvant treatment prior to study enrollment
* Score of < 4 on U.S. Household Food Security Survey Module: Six-Item Short Form OR if score >5, have clearance from dietitian

Exclusion Criteria:

* History of cytotoxic chemotherapy ≤12 months prior to rectal or breast cancer diagnosis
* Allergic reaction to any of the treatment agents
* Any prior pelvic radiotherapy
* Currently active second malignancy other than non-melanoma skin cancers or cervical carcinoma in situ
* History of GI perforation ≤12 months prior to enrollment
* History of predisposing colonic or small bowel disorders with severe or rapidly worsening symptoms (not related to current cancer symptoms)
* Receiving any parenteral nutrition or enteral (tube) feeding or using similar nutritional supplement during the study period
* History of uncontrolled CHF defined as NYHA Class III or greater
* Pre-existing grade ≥3 neuropathy
* Currently participating in or has participated in a study of an investigational agent or investigational device ≤4 weeks of the first dose of treatment
* Unstable psychiatric, sleep, or circadian conditions (common conditions such as sleep apnea and
* depression are acceptable as long as they are stabilized and not rapidly worsening)
* Pregnant or breastfeeding
* Currently perform overnight shift work more than one day/week on average Strictly adhering to a <10-hour eating window on most days
* Known psychiatric or substance misuse disorders that would interfere with adhering to the requirements of the trial

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2029-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Pathological Complete Response (pCR) rate | At completion of neoadjuvant treatment (6 months)
  The pCR will be defined as an absence of residual invasive cancer on hematoxylin and eosin evaluation of the complete resected rectal specimen and all sampled regional lymph nodes. It will be treated as a binary variable.
Treatment-related toxicity | From enrollment till completion of neoadjuvant treatment (6 months)
  The Patient Reported Outcome-Common Terminology Criteria for Adverse Events (PRO-CTCAE v.5) measurement system will be used to measure treatment-related toxicities. The PRO-CTCAE will be administered on a weekly basis throughout the intervention and will calculate the average over all items for each time point. Surveys will be timed relative to the start of each oncologic treatment segment.

SECONDARY OUTCOMES:
Clinical Complete Response (cCR) | At completion of neoadjuvant treatment (6 months)
  A cCR will be defined as the clinical absence of residual disease on physical examination, endoscopic examination, and/or repeat MRI imaging following completion of total neoadjuvant treatment.
Tumor volume | From baseline to surgery (approximately 6 months)
  Standard of care CT and MRI images will be obtained at the time of diagnosis for staging. A repeat standard of care MRI imaging may be obtained prior to surgery to assess response to neoadjuvant therapy and to guide clinical and surgical management. Researchers will obtain routine clinical restaging scans from participants and use them to estimate changes in tumor volume between the two time points.
Objective response rate (ORR) | At the time of surgery (approximately 6 months/days)
  The ORR is defined as the percentage of people who have a partial response (defined as a decrease in tumor volume) or a complete response to treatment between enrollment and surgery.
Adherence | From enrollment till completion of study participation (6 months)
  Adherence will be defined as at least 70% of the daily regimen followed (for example, eating <8 hours for 6 or more days per week on average during the 6-month treatment period). Participants will be asked to self-report their adherence using a weekly survey, which asks participants to record the time they start and finish eating each day and to document any reasons for non-adherence.
Health-related quality of life (HR-QOL) | From enrollment till completion of neoadjuvant treatment (6 months)
  We will use the widely-used and validated European Organization for Research and Treatment of Cancer Quality of Life (QOL) core questionnaire C30 (EORTC QLQ-C30) and the colorectal-cancer specific questionnaire (EORTC CR29). For this study, we focus on highly prevalent rectal cancer treatment-related symptoms, including fatigue, insomnia, pain and bowel-related items (stool frequency, flatulence, and fecal incontinence).
Neoadjuvant rectal (NAR) score | At completion of neoadjuvant treatment (6 months)
  The NAR score is a validated surrogate endpoint for oncologic outcomes used in rectal cancer clinical trials. It takes as input the pathologic nodal status and the clinical and pathologic T-stage.
Provider-reported adverse events | From enrollment till completion of neoadjuvant treatment (6 months)
  As secondary measures of toxicity, researchers will collect provider-reported adverse event data. Researchers will analyze the incidence of grade 3-4 toxicities and calculate the aggregated Toxicity Index (TI). The TI accounts for the frequency and cumulative burden of all toxicities during the treatment period.
Progression-free survival (PFS) | 12- and 24 months post completion of neoadjuvant treatment and surgery
Relapse-free survival (RFS) | 12- and 24 months post completion of neoadjuvant treatment and surgery
Overall survival (OS) | 12- and 24 months post completion of neoadjuvant treatment and surgery

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Thomas, MD, Principal Investigator — Alaska Native Tribal Health Consortium (ANTHC); Jane Figueiredo, PhD, M.Sc., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Alaska Native Medical Center (ANMC), Anchorage, Alaska, United States

IPD SHARING:
Plan to Share IPD: No